CLINICAL TRIAL: NCT05830994
Title: Randomized Sham-controlled Trial Investigating Efficacy of Gastric Peroral Endoscopic Myotomy in Treatment of Diabetic Gastroparesis
Brief Title: Trial Investigating Efficacy of G-POEM
Acronym: G-POEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Zealand University Hospital (Other); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Melina Svraka Hansen, Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJ-981
Record Dates: First submitted 2023-04-12; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Gastroparesis With Diabetes Mellitus
Keywords: gastroparesis; G-POEM; gastric peroral endoscopic myotomy; technetium-scintigraphy
MeSH Terms: conditions — Gastroparesis | interventions — Pyloromyotomy; salicylhydroxamic acid; Endoscopy; Histocompatibility Testing

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to either the group receiving G-POEM or to the control group where a sham procedure consisting of a gastroscopy with biopsy during general anaesthesia will be done. The randomization will be carried out per-operatively. A computer-generated bloc randomization with sizes of four will be applied.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and researchers will be blinded to allocation in the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-POEM procedure (Active Comparator): Gastric peroral endoscopic myotomy
  Interventions: Procedure: G-POEM
- Sham procedure (Placebo Comparator): sham endsocopy with biopsy
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: G-POEM — An Endoscopic submucosal tunnel is formed and extended to the first part of the duodenum, followed by a pyloromyotomy, beginning approximately two centimetres proximal to the pylorus and ending in the first part of duodenum.
  Arms: G-POEM procedure
Procedure: Sham — Endoscopy is performed and tissue samples are collected from fundus and antrum as part of the Sham procedure
  Other Names: Endoscopy with tissue sample
  Arms: Sham procedure

SUMMARY:
The goal of this randomized sham-controlled trial is to ivestigate efficacy and safety of G-POEM in treatment of diabetic gastroparesis and explore impact of G-POEM on glucose metabolism and incretine hormones.

DETAILED DESCRIPTION:
Study Design The study is a single-centre double-blinded sham-controlled randomized trial. All patients have the same baseline characterization. Patients and researchers will be blinded to allocation in trial. Before randomization patients will have an additional meal test performed addressing metabolic characterization of the incretine hormones at baseline. Patients will afterwards be allocated to either the group receiving G-POEM or to the control group where a sham procedure consisting of a gastroscopy with biopsy during general anaesthesia will be done. The randomization will be carried out per-operatively. A computer-generated bloc randomization with sizes of four will be applied. The study will consist of 5 study visits, with a follow-up of 90 days after procedure. Symptoms and adverse event will be monitored 7, 30, and 90 days after intervention. During the 90-day follow-up all primary and secondary outcome will be reassessed.

G-POEM procedure is carried out in general anaesthesia in the operating theatre at the Department of Surgery, Hvidovre Hospital. Procedures will be performed by experienced surgeons from the Gastro Unit at Hvidovre Hospital,who postoperatively will have no contact with the research team or study participants. Patients will receive the same care during hospitalization.

Patients allocated to sham procedure will have 4 mucosa biopsies from antrum. All biopsies will be handled with formalin and transported to Zealand University Hospital. Here they will be formalin fixed paraffin-embedded and kept in a biobank.

ELIGIBILITY:
Inclusion Criteria:

* The ability to give signed written informed consent,
* Patients with diabetes and gastroparesis,
* Age >18 years,
* Gastroparesis is diagnosed with technetium-scintigraphy,
* Normal gastroscopy,

Exclusion Criteria:

* Ongoing cancer treatment or other concurrent illness that will make the patient unable to attend the study on the discretion of the investigator,
* Recent gastrointestinal surgery,
* Active duodenal/gastric ulcer disease,
* Diseases in the ventricle or previously complicated upper abdominal surgery,
* Previous bariatric surgery,
* Pregnancy or breastfeeding,
* Parkinson disease,
* Persons who, in the judgement of the investigator, may be unable to follow the protocol, Use of metoclopramide, domperidone, prucalopride, ghrelin, macrolide antibiotics (eg, azithromycin, clarithromycin, erythromycin) during study period.
* drugs with an anti-cholinergic mechanism,
* Use of motility slowing agents: anticholinergic agents, calcium channel blockers, TCA, GLP-1 analogs, Lithium, diphenhydramin, glucagon, dopamine agonists, progesterone, L-dopa, calcitonine, octreotide, interferon alfa, sucralsulfate,
* botulinum toxin injections (eg, Botox®) by pyloric injection less than 4 months prior to procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in gastric emptying | 90 days after intervention
  assessed by technetium scintigraphy

SECONDARY OUTCOMES:
Changes in gastroparesis cardinal symptom index (GCSI) | 7, 30 and 90 days after intervention.
  patient-rated gastroparesis cardinal symptom index score for gastroparesis-related symptoms (naseau, vomiting, early satiety, postprandial fulness, upper abdominal pain). Range from 0-none to 5-very servere.
Changes in Plasma glucose | 90 days after intervention.
  concentration of plasma glucose in mmol/L
Changes in postprandial incretinhormones | 90 days after intervention.
  gastrin, CCK, GIP, GLP-1, GLP-2, glucagon, ghrelin, pancreatic polypeptide (PP)
Concentration of C-peptide in pmol/L | 90 days after intervention.
  Concentration of C-peptide in pmol/L
Changes in continuous glucose | 90 days after intervention.
  Measure of 10-days interstitial glucose levels with a Dexcom monitor device attached to the abdominal skin
Incidence of Treatment-Emergent Adverse Events rated by the ASGE lexicon for adverse events | 7,30 and 90 days
  rate and severity of adverse events rated by the ASGE lexicon for adverse events

CONTACTS AND LOCATIONS:
Overall Officials: John G Karstensen, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Melina Svraka Hansen, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No